CLINICAL TRIAL: NCT05492773
Title: Evaluating the Efficacy of Micro-Osteoperforations Technique on the Orthodontic Tooth Movement Acceleration of Dental Crowding Cases Treated With Clear Aligners: A Randomized Controlled Clinical Trial
Brief Title: Evaluating the Efficacy of Micro-Osteoperforations Technique on the Orthodontic Tooth Movement Acceleration in Moderate Mandibular Anterior Crowding Cases Treated With Clear Aligners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University -Ortho
Record Dates: First submitted 2022-07-29; First posted 2022-08-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micro-osteoperforations (Experimental): Experimental: Micro-Osteoperforations Technique(MOPs) Experimental: Micro-Osteoperforations Technique(MOPs) Surgery will be performed to the lower anterior bony segment of the lower jaw in order to accelerate tooth movement.
  Interventions: Device: Micro-osteoperforations Technique
- Clear aligner (Experimental): Traditional treatment The patients in this group will be receive treatment with the traditional clear aligners technique without any surgical procedure.
  Interventions: Device: Active comparater

INTERVENTIONS:
Device: Micro-osteoperforations Technique — Micro-Osteoperforations Technique (MOPs) Surgery will be performed to the lower anterior bony segment of the lower jaw in order to accelerate tooth movement.
  Arms: Micro-osteoperforations
Device: Active comparater — Active Comparator: Traditional treatment The patients in this group will be receive treatment with the traditional clear aligners technique without any surgical procedure.
  Arms: Clear aligner

SUMMARY:
Patients with moderate mandibular anterior crowding will be treated in this study. The efficacy of micro-osteoperforations technique by special drill in accelerating orthodontic tooth movement during clear aligners therapy will be assessed along with patient's pain and satisfaction.

There are two groups:

1. a group of patients in which participants will be received treatment with the traditional clear aligners technique in addition to a micro-osteoperforations technique.
2. a group of patients in which participants will be received treatment with the traditional clear aligners technique alone

DETAILED DESCRIPTION:
Dental crowding is one of the most common orthodontic problems in adults as it was found that 80% of adults had crowding in the lower incisors area.

Although many adults need orthodontic treatment, they do not like and sometimes refuse to apply fixed orthodontic devices, so the emergence of Clear Aligners Technique (CAT) where the aesthetic aspect is one of the most important characteristics of this technique which can alleviate the response and anxiety of adult patients related to orthodontic treatment, its approach relies on the use of a series of clear aligners that slowly move each tooth into the desired position.

But the strict protocol that requires wearing each aligner 22 hours a day leads to poor patient compliance with it during the treatment period, so many clinical and laboratory attempts have been made to find different methods that achieve faster results and reduce the extent of orthodontic treatment, and among all the previous methods, the surgical approach is the most clinically used and the most tested with known expectations and stable results.

Although these surgical methods have proven effective, they are considered aggressive in nature as they require lifting of full-thickness buccal and lingual flaps with extensive removal of the buccal and lingual cortical bone, in addition to the fact that they may face rejection of the patient due to anxiety and fear of pain and undergo surgery, patients are usually not open toward ideas involving surgery unless it is the only option to obtain a good bite.

Hence, the interest has increased dramatically in recent years to develop conservative surgical techniques that provide similar clinical efficacy with minimal trauma and greater acceptance by patients. One of these techniques is the micro-osteoperforations technique, which is ideal for adult patients who have limited time and wish to finish their treatment as quickly as possible.

To date, no randomized controlled trial (RCT) has been conducted to study the effects of micro-osteoperforations Technique on the duration of orthodontic treatment along with patient's pain and satisfaction during clear aligner therapy (CAT) in moderate mandibular anterior crowding cases which are one of the most common types of malocclusions.

The current study will have two parallel arms as following:

Group 1 (the intervention group): patients in which participants will be received treatment with the traditional clear aligners technique in addition to a micro-osteoperforations technique.

Group 2 (the control group): patients in which participants will be received treatment with the traditional clear aligners technique alone.

In the intervention and control groups: patients will change aligners depending on the fit of the new aligner.

In the intervention group:

On the placing day of the initial clear aligner, special drill (1 mm in diameter and 10 mm in length) were used to perform the MOPs procedure in the intervention group. Buccal transmucosal MOPs were performed between mandibular canine and first mandibular premolar bilaterally and between mandibular canine and lateral incisor bilaterally and between mandibular lateral incisor and central incisor bilaterally and between central incisors in the midline on labial aspect of mandible.

Two MOPs at each site were performed, first perforation will be performed at a distance of 2mm from free gingival margin and second perforation will be performed 2mm from the first one in a vertical line (which will measure using customized length guides on special drill), making a total of fourteen MOPs.

The depth of perforation will be 1mm in buccal cortical bone (which will measure using customized depth guides on special drill).

ELIGIBILITY:
Inclusion Criteria:

* Completion of permanent dentition (except third molars)
* Moderate crowding (4-6 mm according to Little's index)
* Absence of medications intake that interferes with pain perception for at least one week before the beginning of the treatment
* Number of aligners ≥ 8 aligners.

Exclusion Criteria:

* • Systematic diseases that could affect bone and tooth movement and no contraindication avoid oral surgery

  * Medical conditions that affect tooth movement (Corticosteroid, NSAIDs)
  * Patients had previous orthodontic treatments
  * Poor oral hygiene or concurrent periodontal disease

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-06-10 (Estimated); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Change in Little's Index of Irregularity | T0: immediately before the start of orthodontic treatment; T1: after one month; T2: after two months; T3: after 5 months when Little's Index of Irregularity less than 1 mm and final aligner does not apply any pressure
  The irregularity of the lower incisors is calculated by measuring the amount of deviations of the anatomic contact points between the six anterior teeth in the horizontal direction in mm, since the sum of these measurements represents the value of the index (Little, 1975). When the sum of these deviations is less than 3 mm, this indicates that the teeth are slightly crowded. When the sum is greater than 10 mm, this indicated very severe crowding. The ordinary orthodontic treatment aims to keep this Index less than 1 mm at the end of treatment.
Overall treatment Time | After 5 months when Little's Index of Irregularity less than 1 mm and final aligner will be properly fitting and does not apply any pressure on the teeth with absolute ease of placing and removing it from the teeth,
  the overall time required to complete the treatment was calculated by calculating the number of days between (To) and (T3).

SECONDARY OUTCOMES:
Change in the levels of pain | 4 ,12,24,48 hours following the onset of orthodontic treatment
  Pain is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of pain being experienced. The left end of the line refers to no pain (VAS=0) where the right end refers to maximum (unimaginable) pain (VAS=100). The level of pain is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the pain.
Satisfaction using VAS | After 5 months when Little's Index of Irregularity less than 1 mm and final aligner will be properly fitting and does not apply any pressure on the teeth with absolute ease of placing and removing it
  satisfaction is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of satisfaction. The left end of the line refers to no satisfaction (VAS=0) where the right end refers to maximum satisfaction (VAS=100). The level of satisfaction is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the satisfaction.
Satisfaction with the ease of the procedure | After 5 months when Little's Index of Irregularity less than 1 mm and final aligner will be properly fitting and does not apply any pressure on the teeth with absolute ease of placing and removing it from the teeth,
  is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of ease. The left end of the line refers to no ease (VAS=0) where the right end refers to maximum ease (VAS=100). The grade of ease is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the ease of the procedure.
Satisfaction through acceptability of the procedure | After 5 months when Little's Index of Irregularity less than 1 mm and final aligner will be properly fitting and does not apply any pressure on the teeth with absolute ease of placing and removing it from the teeth,]
  Patients in micro-Osteoperforations group were asked about possibility of repeating the procedure, and they answered using a two-point scale (1. Yes or 2. No).
Satisfaction through recommending the procedure | After 5 months when Little's Index of Irregularity less than 1 mm and final aligner will be properly fitting and does not apply any pressure on the teeth with absolute ease of placing and removing it from the teeth
  Recommendation to a friend: Patients in micro-Osteoperforations group were asked about making recommendation to a friend, and they answered using a two-point scale (1. Yes or 2. No).

CONTACTS AND LOCATIONS:
Overall Officials: Zouha Barram, Principal Investigator — Hama University; Rabab AlSabbag, Professor, Study Director — Hama University
Locations (1):
- Hama University, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] Al-Khalifa KS, Baeshen HA. Micro-osteoperforations and Its Effect on the Rate of Tooth Movement: A Systematic Review. Eur J Dent. 2021 Feb;15(1):158-167. doi: 10.1055/s-0040-1713955. Epub 2020 Jul 1. PMID 32610360
- [Background] Al-Dboush R, Esfahani AN, El-Bialy T. Impact of photobiomodulation and low-intensity pulsed ultrasound adjunctive interventions on orthodontic treatment duration during clear aligner therapy. Angle Orthod. 2021 Sep 1;91(5):619-625. doi: 10.2319/112420-956.1. PMID 34407180
- [Background] Monnerat C, Restle L, Mucha JN. Tomographic mapping of mandibular interradicular spaces for placement of orthodontic mini-implants. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):428.e1-9; discussion 428-9. doi: 10.1016/j.ajodo.2008.12.003. PMID 19361724
- [Background] Purmal K, Alam MK, Pohchi A, Abdul Razak NH. 3D mapping of safe and danger zones in the maxilla and mandible for the placement of intermaxillary fixation screws. PLoS One. 2013 Dec 19;8(12):e84202. doi: 10.1371/journal.pone.0084202. eCollection 2013. PMID 24367643
- [Background] Sadek MM, Sabet NE, Hassan IT. Three-dimensional mapping of cortical bone thickness in subjects with different vertical facial dimensions. Prog Orthod. 2016 Dec;17(1):32. doi: 10.1186/s40510-016-0145-x. Epub 2016 Oct 17. PMID 27667817
- [Background] Tepedino M, Cattaneo PM, Masedu F, Chimenti C. Average interradicular sites for miniscrew insertion: should dental crowding be considered? Dental Press J Orthod. 2017 Sep-Oct;22(5):90-97. doi: 10.1590/2177-6709.22.5.090-097.oar. PMID 29160349
- [Background] Wang Y, Shi Q, Wang F. Optimal Implantation Site of Orthodontic Micro-Screws in the Mandibular Anterior Region Based on CBCT. Front Physiol. 2021 May 20;12:630859. doi: 10.3389/fphys.2021.630859. eCollection 2021. PMID 34093218